CLINICAL TRIAL: NCT00629811
Title: A Double-Blind, Placebo-Controlled, Randomised Dose Ranging Trial to Investigate the Efficacy of Two Different Dosing Regimens of Avotermin (Juvista) in the Improvement of Scar Appearance When Applied to Approximated Wound Margins in Healthy Volunteers.
Brief Title: Improvement in Scar Appearance Following Injection of Avotermin (Juvista) Into Skin Incisions Made in Healthy Men and Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Mr Mark Cooper, Senior Vice President of Clinical Operations, Renovo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RN1001-0036
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-02

CONDITIONS: Cicatrix
Keywords: Cicatrix; Scar; TGFβ3; Avotermin; Juvista; RN1001
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human; Transforming Growth Factor beta3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Avotermin (Juvista) — Intradermal avotermin administered to four wound sites per subject, one wound site per anatomically matched pair, according to the subject's assigned dose group:
  * Group 1: avotermin concentrations of 5, 50, 200 and 500ng per 100μL per linear cm of wound site (pre-wounding, Day 0) and 100μL per linear cm of wound margin (post-wounding, Day 1)
  * Group 2: avotermin concentrations of 5, 50, 200 and 500ng per 100μL per linear cm of wound site (pre-wounding, Day 0) and 100μL per linear cm of wound margin (post-wounding, Day 0)
  Each subject received four doses of active drug at concentrations of 5, 50, 200 and 500ng per 100μL per linear cm of wound site, one dose to one wound site per anatomically matched pair of wounds.
  Other Names: Juvista, RN1001, transforming-growth factor beta 3, TGFβ3
Drug: Placebo — Reference therapy was Placebo (vehicle). On Day 0, the four sites randomised to receive Placebo were administered with a 100μL intradermal injection of Placebo.
  Subjects in Group 2 were dosed again on Day 0 at 10 to 30 minutes after wound closure.
  Subjects in Group 1 were dosed again on Day 1 at 24 (+/-4) hours after initial administration of drug.

SUMMARY:
This is a single-centre, double-blind, Placebo-controlled, randomised trial. Trial subjects received four 1cm incisional wounds on the inner aspect of each upper arm (eight in total), giving four pairs of anatomically matched wound sites per subject. Each subject acted as their own control. One site from each anatomical wound pair was randomly treated with intradermally administered avotermin (Juvista:100μL per linear cm of wound site pre-operatively and 100μL per linear cm of wound margin post-wounding on Day 0 or Day 1, 400μL per wound site) while the second site was a paired control, treated with Placebo (100μL per linear cm of wound site pre-operatively and 100μL per linear cm of wound margin post-wounding on Day 0 or Day 1, 400μL per wound site). Wound margins for injection were defined as extending 0.5cm from either end of the incision. Four doses of avotermin (Juvista) were administered to each subject: 5ng, 50ng, 200ng and 500ng/100μL per linear cm; one dose to one wound site per anatomically matched pair of wounds. The second wound site from each anatomically matched pair of wounds was dosed with placebo. Allocation of treatment to wound-site pairs was randomised and double blinded.

Primary objective To determine the optimal concentration and dose regimen of Juvista for the improvement of the resultant scar when applied to the approximated wound margins of male and female subjects following surgical incisions.

Secondary objective To assess the safety and tolerance of Juvista when applied to the approximated wound margins of male and female subjects following surgical incisions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-85 years who have given written informed consent.
* Subjects with a body mass index within 15-35 kg/m2 (Quetelet's index).

Exclusion Criteria:

* Subjects with history or evidence of keloid scarring.
* Subjects with tattoos or previous scars within 3cm of the area to be incised.
* Subjects who had surgery in the area to be incised within one year of the first dosing day.
* Subjects with history of a bleeding disorder or who were receiving anti-coagulant or anti-platelet therapy.
* Subjects with evidence of any past or present clinically significant disease that may affect the endpoints of the trial.
* Subjects with a clinically significant skin disorder that was chronic or currently active.
* Subjects with any clinically significant medical condition or history that would impair wound healing.
* Subjects with history of hypersensitivity to any of the drugs or dressings used in this trial.
* Subjects taking, or who have taken, any investigational product or who had participated in a clinical trial in the three months prior to first trial dose administration.
* Subjects taking regular, continuous, oral corticosteroid therapy.
* Subjects undergoing investigations or changes in management for an existing medical condition.
* Subjects with a history of drug abuse, or with a positive drugs of abuse test for cocaine, amphetamines, methamphetamines, opiates or benzodiazepines during the screening period.
* Subjects who, in the opinion of the investigator, were unlikely to complete the trial for whatever reason.
* Subjects who had any clinically significant neurological impairment or disease.
* Subjects with any active infection.
* Subjects who are pregnant or lactating.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To determine the optimal concentration and dose regimen of avotermim (Juvista) for the improvement of the resultant scar when applied to the approximated wound margins of male and female subjects following surgical incisions. | Post surgery: week 6 to Month 7

SECONDARY OUTCOMES:
To assess the safety and tolerance of avotermin (Juvista) when applied to the approximated wound margins of male and female subjects following surgical incisions. | Day 0 (surgery) to Month 7 post surgery

CONTACTS AND LOCATIONS:
Overall Officials: James Bush, MBChB, Principal Investigator — Renovo
Locations (1):
- Clinical Trials Unit, Renovo, Manchester, United Kingdom

REFERENCES:
- [Derived] Ferguson MW, Duncan J, Bond J, Bush J, Durani P, So K, Taylor L, Chantrey J, Mason T, James G, Laverty H, Occleston NL, Sattar A, Ludlow A, O'Kane S. Prophylactic administration of avotermin for improvement of skin scarring: three double-blind, placebo-controlled, phase I/II studies. Lancet. 2009 Apr 11;373(9671):1264-74. doi: 10.1016/S0140-6736(09)60322-6. PMID 19362676